CLINICAL TRIAL: NCT03894696
Title: Frequency of Anxiety and Depression in Chronic Hepatitis C Patients Recieving Direct-Acting Antiviral Agents.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Khaled Mostafa Mohamed, resident at gastroenterology and tropical medicine -Assiut university, Assiut University
Other Study IDs: DAAs and psychiatry
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Direct Acting Antivirals — follow up chronic HCV patients recieving DAAs to detect anxiety and depression

SUMMARY:
The primary objective of this study is to prospectively analyse psychiatric outcomes, specifically depression and anxiety in patients with hepatitis C virus infection who are initiated on DAA therapy (sofosbuvir based regimen).

DETAILED DESCRIPTION:
Hepatitis C is a major cause of chronic liver disease worldwide with an estimated 71 million people infected in 2015 and approximately 1.75 million new infections each year .

Egypt had high burden of liver disease from viral hepatitis , and near to 15% of the adult population had HCV seropositivity and more than 4 million persons had also viraemia .

The discovery of direct-acting antiviral agents (DAAs) has dramatically changed HCV treatment by increasing the cure rate and decreasing the duration of therapy .The current generation of DAAs (e.g., daclatasvir [DCV], sofosbuvir [SOF], simeprevir [SIM] and ledipasvir [LDV]) is used without IFN .

The approval of direct - acting antiviral (DAA) agents revolutionized HCV treatment and allowed for non-IFN-a-based regimens. Psychiatric and psychosocial contraindications to treatment are reduced due to shorter duration of therapy and improved side effect profiles . Also, the favorable side effect profiles of DAA agents (less fatigue and blood dyscrasias) lead to high adherence rates of 96.2%, compared to 84.3% and 77.6% in IFN-free RBV-containing regimens and IFN- and RBV containing regimen respectively .

Sofosbuvir and daclatasvir are new direct acting antivirals (DAAs) which are tolerable and safe. Daclatasvir is a first-in-class HCV NS5A replication complex inhibitor with pangenotypic activity and can be used once-daily. Sofosbuvir is an orally administered HCV nucleotide polymerase NS5B inhibitor. It is given once daily with a good safety profile . The sofosbuvir and daclatasvir combination is associated with a high rate of SVR in difficult-to-treat patients infected with genotype 1 or 4. Addition of ribavirin increases the SVR rate in cirrhotic and treatment-experienced patients .

Mental illness are significantly higher in chronic HCV patients than in the general population, with depression, schizophrenia, and bipolar disorder occurring at 25%, 3.9%, and 2.6% respectively . HCV infection lead to psychiatric symptoms by inflammatory routes, direct brain neurotoxicity, metabolic and neurotransmitter pathway derangement and immune-mediated responses . Currently, the extent of psychiatric effects attributed to DAA agents is unclear; however, it is less than IFN-containing regimens . Though data suggests that DAAs confer a minimal risk of psychiatric adverse effects compared to IFN-based regimens; there is a paucity of data specifically adressing neuropsychiatric complications of these drugs. In addition, it is unclear whether DAA therapy may exacerbate mood symptoms in patients with prior psychiatric history .

ELIGIBILITY:
Inclusion Criteria:

18 years and older Chronic Hepatitis C infection Naive patients who will start a 12-week DAA therapy Acceptance to share in study

Exclusion Criteria:

Recieving antipsychotic . Previous failure of DAA agents. Significant life-threatening diseases HCV related liver cirrhosis. Non HCV related liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the inclusion criteria will attend the hepatitis outpatient clinic of Al-Rajhi Liver Hospital. Selected patients will be followed up for 6 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
frequency of anxiety and depression in chronic HCV patients recieving DAAs. | 6 months .
  to detect occurance of psychatric disorders specifically anxiety and depression in chronic HCV patients treated with DAAs ( sofosbuvir based regimens).

REFERENCES:
- [Background] Sockalingam S, Sheehan K, Feld JJ, Shah H. Psychiatric care during hepatitis C treatment: the changing role of psychiatrists in the era of direct-acting antivirals. Am J Psychiatry. 2015 Jun;172(6):512-6. doi: 10.1176/appi.ajp.2015.14081041. No abstract available. PMID 26029803
- [Background] Tang LS, Masur J, Sims Z, Nelson A, Osinusi A, Kohli A, Kattakuzhy S, Polis M, Kottilil S. Safe and effective sofosbuvir-based therapy in patients with mental health disease on hepatitis C virus treatment. World J Hepatol. 2016 Nov 8;8(31):1318-1326. doi: 10.4254/wjh.v8.i31.1318. PMID 27872683
- [Background] Rowan PJ, Bhulani N. Psychosocial assessment and monitoring in the new era of non-interferon-alpha hepatitis C virus treatments. World J Hepatol. 2015 Sep 8;7(19):2209-13. doi: 10.4254/wjh.v7.i19.2209. PMID 26380046
- [Background] Younossi ZM, Stepanova M, Henry L, Nader F, Younossi Y, Hunt S. Adherence to treatment of chronic hepatitis C: from interferon containing regimens to interferon and ribavirin free regimens. Medicine (Baltimore). 2016 Jul;95(28):e4151. doi: 10.1097/MD.0000000000004151. PMID 27428205
- [Background] Wu JY, Shadbolt B, Teoh N, Blunn A, To C, Rodriguez-Morales I, Chitturi S, Kaye G, Rodrigo K, Farrell G. Influence of psychiatric diagnosis on treatment uptake and interferon side effects in patients with hepatitis C. J Gastroenterol Hepatol. 2014 Jun;29(6):1258-64. doi: 10.1111/jgh.12515. PMID 24955454
- [Background] Sockalingam S, Tseng A, Giguere P, Wong D. Psychiatric treatment considerations with direct acting antivirals in hepatitis C. BMC Gastroenterol. 2013 May 14;13:86. doi: 10.1186/1471-230X-13-86. PMID 23672254
- [Background] Jacobson IM, Dore GJ, Foster GR, Fried MW, Radu M, Rafalsky VV, Moroz L, Craxi A, Peeters M, Lenz O, Ouwerkerk-Mahadevan S, De La Rosa G, Kalmeijer R, Scott J, Sinha R, Beumont-Mauviel M. Simeprevir with pegylated interferon alfa 2a plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 infection (QUEST-1): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2014 Aug 2;384(9941):403-13. doi: 10.1016/S0140-6736(14)60494-3. Epub 2014 Jun 4. PMID 24907225
- [Background] Tully DC, Hjerrild S, Leutscher PD, Renvillard SG, Ogilvie CB, Bean DJ, Videbech P, Allen TM, McKeating JA, Fletcher NF. Deep sequencing of hepatitis C virus reveals genetic compartmentalization in cerebrospinal fluid from cognitively impaired patients. Liver Int. 2016 Oct;36(10):1418-24. doi: 10.1111/liv.13134. Epub 2016 Apr 26. PMID 27045383
- [Background] Pol S, Corouge M, Vallet-Pichard A. Daclatasvir-sofosbuvir combination therapy with or without ribavirin for hepatitis C virus infection: from the clinical trials to real life. Hepat Med. 2016 Mar 4;8:21-6. doi: 10.2147/HMER.S62014. eCollection 2016. PMID 27019602
- [Background] Sofia MJ, Bao D, Chang W, Du J, Nagarathnam D, Rachakonda S, Reddy PG, Ross BS, Wang P, Zhang HR, Bansal S, Espiritu C, Keilman M, Lam AM, Steuer HM, Niu C, Otto MJ, Furman PA. Discovery of a beta-d-2'-deoxy-2'-alpha-fluoro-2'-beta-C-methyluridine nucleotide prodrug (PSI-7977) for the treatment of hepatitis C virus. J Med Chem. 2010 Oct 14;53(19):7202-18. doi: 10.1021/jm100863x. PMID 20845908
- [Background] Gao M, Nettles RE, Belema M, Snyder LB, Nguyen VN, Fridell RA, Serrano-Wu MH, Langley DR, Sun JH, O'Boyle DR 2nd, Lemm JA, Wang C, Knipe JO, Chien C, Colonno RJ, Grasela DM, Meanwell NA, Hamann LG. Chemical genetics strategy identifies an HCV NS5A inhibitor with a potent clinical effect. Nature. 2010 May 6;465(7294):96-100. doi: 10.1038/nature08960. Epub 2010 Apr 21. PMID 20410884
- [Background] Coppola N, Zampino R, Bellini G, Stanzione M, Capoluongo N, Marrone A, Macera M, Pasquale G, Boemio A, Maione S, Adinolfi LE, Del Giudice EM, Sagnelli E, Rossi F. The impact of the CB2-63 polymorphism on the histological presentation of chronic hepatitis B. Clin Microbiol Infect. 2015 Jun;21(6):609.e1-4. doi: 10.1016/j.cmi.2015.02.021. Epub 2015 Mar 5. PMID 25749560
- [Background] Banerjee D, Reddy KR. Review article: safety and tolerability of direct-acting anti-viral agents in the new era of hepatitis C therapy. Aliment Pharmacol Ther. 2016 Mar;43(6):674-96. doi: 10.1111/apt.13514. Epub 2016 Jan 20. PMID 26787287
- [Background] Kandeel A, Genedy M, El-Refai S, Funk AL, Fontanet A, Talaat M. The prevalence of hepatitis C virus infection in Egypt 2015: implications for future policy on prevention and treatment. Liver Int. 2017 Jan;37(1):45-53. doi: 10.1111/liv.13186. Epub 2016 Jun 30. PMID 27275625
- [Background] Stanaway JD, Flaxman AD, Naghavi M, Fitzmaurice C, Vos T, Abubakar I, Abu-Raddad LJ, Assadi R, Bhala N, Cowie B, Forouzanfour MH, Groeger J, Hanafiah KM, Jacobsen KH, James SL, MacLachlan J, Malekzadeh R, Martin NK, Mokdad AA, Mokdad AH, Murray CJL, Plass D, Rana S, Rein DB, Richardus JH, Sanabria J, Saylan M, Shahraz S, So S, Vlassov VV, Weiderpass E, Wiersma ST, Younis M, Yu C, El Sayed Zaki M, Cooke GS. The global burden of viral hepatitis from 1990 to 2013: findings from the Global Burden of Disease Study 2013. Lancet. 2016 Sep 10;388(10049):1081-1088. doi: 10.1016/S0140-6736(16)30579-7. Epub 2016 Jul 7. PMID 27394647
- [Background] World Health Organization. Hepatitis C. WHO fact Sheet 164 2017. [http://www.who.int/mediacentre/factsheets/fs164/en/].
- [Background] Younossi Z, Henry L. Systematic review: patient-reported outcomes in chronic hepatitis C--the impact of liver disease and new treatment regimens. Aliment Pharmacol Ther. 2015 Mar;41(6):497-520. doi: 10.1111/apt.13090. Epub 2015 Jan 23. PMID 25616122